CLINICAL TRIAL: NCT04471207
Title: Intelligent Biometrics to Optimize Prolonged Exposure for PTSD
Brief Title: Clinical Trial Intelligent Biometrics for PTSD - Clinical Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Zeriscope (Industry)
Responsible Party: Principal Investigator, Sudie E. Back, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00094890
Record Dates: First submitted 2020-04-14; First posted 2020-07-15 (Actual); Results first posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: PTSD
Keywords: PTSD; Military; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intelligent Biometrics - Prolonged Exposure (Therapist Guided). (Experimental): In the therapist-guided group, Study Therapists will virtually accompany patients during IVEs and use actionable biometric and subjective data during in vivo exposures (IVEs) (galvanic skin response [GSR], heart rate [HR], and subjective units of distress [SUDS]) to modify the assignments in real-time.
  All participants receive at least 10 sessions of prolonged exposure therapy for posttraumatic stress disorder.
  Interventions: Device: Therapist Guided Prolonged Exposure with BioWare Device
- Intelligent Biometrics - Prolonged Exposure (Record Only). (Active Comparator): In the record-only group, passive data collection will be utilized to collect and store biometric and behavioral data for future offline analyses to investigate predictors of outcome.
  All participants receive at least 10 sessions of prolonged exposure therapy for posttraumatic stress disorder.
  Interventions: Device: Record Only Prolonged Exposure with BioWare Device

INTERVENTIONS:
Device: Therapist Guided Prolonged Exposure with BioWare Device — Experimental: Intelligent Biometrics - Prolonged Exposure (therapist guided). In the therapist guided group, Study Therapists will use actionable data during in vivo exposures (IVEs) (galvanic skin response [GSR], heart rate [HR], and subjective units of distress [SUDS]) to modify the assignments in real-time.
  All participants receive at least 10 sessions of prolonged exposure therapy for posttraumatic stress disorder.
  Arms: Intelligent Biometrics - Prolonged Exposure (Therapist Guided).
Device: Record Only Prolonged Exposure with BioWare Device — In the record-only group, passive data collection will be utilized to collect and store biometric and behavioral data for future offline analyses to investigate predictors of outcome.
  All participants receive at least 10 sessions of prolonged exposure therapy for posttraumatic stress disorder.
  Arms: Intelligent Biometrics - Prolonged Exposure (Record Only).

SUMMARY:
Posttraumatic stress disorder (PTSD) is a debilitating mental health condition that increases suicide risk and affects up to 20% of military veterans and 8% of the general population. Prolonged Exposure (PE) is a highly effective behavioral (talk therapy) intervention for PTSD. However, dropout rates are high (25-30%) and an estimated one-third of patients who complete PE still report symptoms of PTSD at the end of treatment. This study directly addresses these limitations by using a clinical trial to evaluate the ability of an innovative technology system to improve PE therapy for veterans with PTSD.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a chronic and debilitating psychiatric condition. Prolonged Exposure (PE) therapy is a highly effective, evidence-based treatment for PTSD; however, dropout rates are high and approximately one-third of patients who complete treatment remain symptomatic. The proposed study will employ a randomized clinical trial (N=40 treatment-seeking veterans with current PTSD) to evaluate the acceptability, feasibility and preliminary efficacy of a technological enhancement (IB-PE), and investigate predictors of outcome by accomplishing the following milestones: (1a) Evaluate ability of IB-PE (therapist guided vs. record only) in reducing PTSD severity from baseline to end of treatment; and (2b) Use a variety of in vivo exposures (IVEs) to identify biometric and behavioral indicators (high heart rate, skin conductance) with high predictive value of treatment response. We will use a technology system of discrete wearables (camera, microphone) to allow therapists to accompany participants during IVEs. The system will pair with a cellular application and record information such as heart rate and skin conductance. This system will also allow the participant to communicate with the study therapist during the guided in vivo exercises.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; any race or ethnicity; aged 18-75 years.
2. U.S. Military veteran, any branch or era.
3. Participants must be able to comprehend English.
4. Participants must meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnostic criteria for current (i.e., past 6 months) posttraumatic stress disorder (PTSD) (assessed via the Clinician Administered PTSD Scale for DSM-5). Subjects may also meet criteria for a mood disorder (except bipolar affective disorder, see Exclusion Criteria) or anxiety disorders (panic disorder, agoraphobia, social phobia, generalized anxiety disorder, or obsessive compulsive disorder). The inclusion of subjects with affective and other anxiety disorders is essential because of the marked frequency of the co-existence of mood and other anxiety disorders among patients with PTSD.
5. Participants taking psychotropic medications will be required to be maintained on a stable dose for at least four weeks before study initiation.

Exclusion Criteria:

1. Participants meeting DSM-5 criteria for a history of or current psychotic or bipolar affective disorders. Those participants will be referred clinically to ensure they have appropriate level of clinical care.
2. Participants meeting DSM-5 criteria for a current (past 6 months) moderate to severe substance use disorder. Those participants will be referred to addiction treatment centers at the Veterans Affairs, Medical University of South Carolina and in the local community. Individuals with mild substance use disorder (SUD) will be included.
3. Participants considered an immediate suicidal or homicidal risk or who are likely to require hospitalization during the course of the study for suicidality. Those participants will be referred clinically for care.
4. Participants on maintenance anxiolytic, antidepressant, or mood stabilizing medications, which have been initiated during the past 4 weeks.
5. Participants enrolled in ongoing evidence-based behavioral therapy for PTSD who are not willing to discontinue these therapies for the duration of the trial. Attendance at therapeutic activities other than study sessions will be closely monitored using the Treatment Services Review.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Saraiya TC, Jarnecke AM, Rothbaum AO, Wangelin B, McTeague LM, Acierno R, Brown DG, Bristol E, Feigl H, Reese M, Cobb AR, Harley B, Adams RJ, Back SE. Technology-enhanced in vivo exposures in Prolonged Exposure for PTSD: A pilot randomized controlled trial. J Psychiatr Res. 2022 Dec;156:467-475. doi: 10.1016/j.jpsychires.2022.10.056. Epub 2022 Nov 1. PMID 36347106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited via online advertisements and clinician referrals. Participants were seen via telehealth due to the coronavirus-2 pandemic (SARS-Cov-2). Of note, the study initially focused on military veterans because of their high levels of posttraumatic stress disorder. However, due to the SARS-Cov-2 pandemic which impacted recruitment goals, the inclusion criteria were expanded to include both civilians and veterans.
Pre-assignment Details: A total of 40 participants were randomized in a 3:1 fashion (Guided, n = 29; Non-Guided, n = 11). One participant was removed from the Non-Guided group due to a medical contraindication, and thus the intent-to-treat (ITT) sample consisted of N = 39 individuals. A total of n = 23 individuals completed at least eight sessions of prolonged exposure therapy and used the BioWare system at least one time and represents the treatment completers or per protocol (PP) sample.
Groups:
- Intelligent Biometrics - Prolonged Exposure (Therapist Guided).: Therapist Guided Prolonged Exposure with BioWare Device: Experimental: Intelligent Biometrics - Prolonged Exposure (therapist guided). In the therapist guided group, Study Therapists use actionable biometric and subjective data during in-vivo exposures (IVEs) (heart rate and subjective units of distress) to modify the assignments in real-time.
  All participants receive prolonged exposure therapy for posttraumatic stress disorder.
- Intelligent Biometrics - Prolonged Exposure (Record Only).: Record Only Prolonged Exposure with BioWare Device: In the record-only group, passive data collection will be utilized to collect and store biometric and behavioral data for future offline analyses to investigate predictors of outcome.
  All participants receive prolonged exposure therapy for posttraumatic stress disorder.
Period: Overall Study
Arm/Group | Intelligent Biometrics - Prolonged Exposure (Therapist Guided). | Intelligent Biometrics - Prolonged Exposure (Record Only).
Started | 29 | 11
Completed | 18 | 5
Not Completed | 11 | 6
Not completed — Lost to Follow-up | 4 | 1
Not completed — Medication Contraindication | 0 | 1
Not completed — Loss of Interest | 2 | 1
Not completed — Unwilling to Discuss Trauma | 1 | 1
Not completed — Scheduling Conflicts | 3 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Unwilling to Use System | 0 | 1

BASELINE CHARACTERISTICS:
Population: 18 years of age or older Able to comprehend English Met diagnostic criteria for current posttraumtic stress disorder (PTSD) Stabilized on any psychotropic medications for at least four weeks prior to study initiation Not at risk for imminent suicidal or homicidal ideation or intent requiring a higher level of care, enrolled in any other evidence based PTSD treatment or implanted with any electronic device (pacemaker, electron pump)
Groups:
- Intelligent Biometrics - Prolonged Exposure (Therapist Guided).: Therapist Guided Prolonged Exposure with BioWare Device: Experimental: Intelligent Biometrics - Prolonged Exposure (therapist guided). In the therapist guided group, Study Therapists use actionable biometric and subjective data during in-vivo exposures (IVEs) (e.g., heart rate and subjective units of distress) to modify the assignments in real-time.
  All participants receive prolonged exposure therapy for posttraumatic stress disorder.
- Total: Total of all reporting groups
Arm/Group | Intelligent Biometrics - Prolonged Exposure (Therapist Guided). | Intelligent Biometrics - Prolonged Exposure (Record Only). | Total
Number analyzed (Participants) | 29 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.34 (15.41) | 48.10 (13.05) | 45.31 (14.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 3 | 18
  Male | 14 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 27 | 9 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 20 | 7 | 27
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Post Traumatic Stress Disorder Symptom Severity - Clinician Rated
Description: Clinician Administered Posttraumatic Stress Disorder (PTSD) Scale (CAPS-5) is a clinician administered assessment for posttraumatic stress symptoms. The assessment is administered at baseline, mid treatment and end of treatment. The CAPS-5 is a 30 item assessment that assesses 20 symptoms of PTSD, with scores ranging from 0-80. Lower scores represent fewer and less sever symptoms of PTSD.
Time Frame: End of treatment (after 10-12 sessions of prolonged exposure). Participants had 24 weeks to complete treatment.
Population: Analysis on treatment completers (completion of at least eight sessions of prolonged exposure and use of BioWare device at least one time.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intelligent Biometrics - Prolonged Exposure (Therapist Guided). | Intelligent Biometrics - Prolonged Exposure (Record Only).
Number analyzed (Participants) | 18 | 5
units on a scale | 25.71 (14.65) | 32.00 (11.64)

2. Primary Outcome: Post Traumatic Stress Disorder Symptom Severity - Self Report
Description: Posttraumatic Checklist for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (PCL-5) is a twenty item assessment for self-reported symptoms of posttraumatic stress symptoms. Assessment was administered at baseline, and weekly through the end of treatment. Each of the twenty items has a score of 0-4. Lower scores represent fewer posttraumatic stress symptoms. Scores range from 0 to 80.
Time Frame: End of treatment (after 10-12 sessions of prolonged exposure). Participants had 24 weeks to complete treatment.
Population: Analysis on treatment completers (completion of at least eight sessions of prolonged exposure and use of Bio Ware device at least one time.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intelligent Biometrics - Prolonged Exposure (Therapist Guided). | Intelligent Biometrics - Prolonged Exposure (Record Only).
Number analyzed (Participants) | 18 | 5
units on a scale | 27.11 (18.56) | 50.80 (17.34)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline through follow up, approximately 4 months.
Groups:
- Intelligent Biometrics - Prolonged Exposure (Therapist Guided).: Therapist Guided Prolonged Exposure with BioWare Device: Experimental: Intelligent Biometrics - Prolonged Exposure (therapist guided). In the therapist-guided group, Study Therapists will virtually accompany patients during in vivo exposures (IVEs) and use actionable biometric and subjective data during IVEs (galvanic skin response [GSR, subjective units of distress [SUDS], and heart rate [HR) to modify the assignments in real-time.
  All participants receive at least 10 sessions of prolonged exposure therapy for posttraumatic stress disorder.
Arm/Group | Intelligent Biometrics - Prolonged Exposure (Therapist Guided). | Intelligent Biometrics - Prolonged Exposure (Record Only).
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/29 | 2/11
Other Adverse Events (participants affected / at risk) | 10/29 | 3/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intelligent Biometrics - Prolonged Exposure (Therapist Guided). (N=29) | Intelligent Biometrics - Prolonged Exposure (Record Only). (N=11)
Intestinal Lymphangiectasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Hospitalization for surgical/medical procedure
Spinal Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Hospitalization for medical/surgical procedure: repair of deterioration of L1 and L5 spinal segments.
Transient Ischemic (Nervous system disorders) | 0 (0) | 1 (1) — Hospitalization after transient ischemic attack (mini stroke)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intelligent Biometrics - Prolonged Exposure (Therapist Guided). (N=29) | Intelligent Biometrics - Prolonged Exposure (Record Only). (N=11)
Headache or Migraine (Nervous system disorders) | 5 (6) | 0 (0)
Cough (Infections and infestations) | 4 (4) | 0 (0)
Gastrointestinal Discomfort (Gastrointestinal disorders) | 3 (6) | 2 (2) — including comiting, stomach virus, nausea and diarrhea
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Fever (Infections and infestations) | 3 (3) | 0 (0)
Pain in Lower Extremities (Musculoskeletal and connective tissue disorders) | 3 (6) | 3 (3) — Pain reported in back, leg, knee

LIMITATIONS AND CAVEATS:
The sample size was small, particularly for the Non-Guided group due to the focus on gaining experience with the clinician-guided IVEs in the Guided group. Thus, power to detect some effects was low, and the findings should be considered preliminary. Guided group also received more attention than Non-Guided group through the delivery of clinician-guided IVEs. This study did not compare between self-guided IVEs with the device and self-guided IVEs without the device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT04471207/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT04471207/ICF_001.pdf